CLINICAL TRIAL: NCT04029662
Title: Comparison of Valsalva Maneuver and Control Technique in Reducing Pain Intensity During Spinal Needle Insertion
Brief Title: Reducing Pain Intensity During Spinal Needle Insertion: Valsalva Maneuver vs. Control Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Alfan Mahdi Nugroho, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes039
Record Dates: First submitted 2019-07-20; First posted 2019-07-23 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Undefined
MeSH Terms: interventions — Valsalva Maneuver

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Valsalva Maneuver (Experimental): Patients who undergo spinal anesthesia and perform Valsalva maneuver to reduce the pain intensity
  Interventions: Behavioral: Valsalva Maneuver
- Group Control (No Intervention): Patients who undergo spinal anesthesia and perform nothing to reduce the pain intensity

INTERVENTIONS:
Behavioral: Valsalva Maneuver — Performing Valsalva maneuver will reduce the pain intensity during spinal needle insertion.
  Arms: Group Valsalva Maneuver

SUMMARY:
This study was aimed to observe the efficacy of Valsalva maneuver in reducing pain intensity during spinal needle insertion.

DETAILED DESCRIPTION:
Spinal anesthesia is one of the regional anesthesia techniques needed to provide motor, sensory, and autonomic blocks specifically for lower limbs by delivering local anesthetics into subarachnoid space. This technique is not difficult to perform and relatively inexpensive. However, spinal anesthesia may cause an intense pain during needle insertion. Valsalva maneuver is an attempt to force expiration by pushing a closed airway, such as covering nose or mouth. This maneuver can lead to anti-nociceptive stimulation and may decrease the pain. Thus, this study was aimed to observe the efficacy of Valsalva maneuver in reducing pain intensity during spinal needle insertion.

ELIGIBILITY:
Inclusion Criteria:

* Elective patients having spinal anesthesia
* Patients with no previous history of spinal anesthesia
* Patients with criteria of American Society of Anaesthesiologist (ASA) I-II
* Patients willing to participate in the study and signing informed consent form

Exclusion Criteria:

* Patients with contraindications of spinal anesthesia
* Patients with difficulty in blowing 30 mmHg for 20 seconds
* Patients having allergic reactions due to local anesthetics and opioid

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Level of Pain Intensity | 15 minutes
  Pain Measurement by Visual Analog Scale or Numeric Rating Scale with Range 1-10

CONTACTS AND LOCATIONS:
Overall Officials: Alfan M Nugroho, MD, Principal Investigator — Indonesia University
Locations (1):
- Indonesia University, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calthorpe N. The history of spinal needles: getting to the point. Anaesthesia. 2004 Dec;59(12):1231-41. doi: 10.1111/j.1365-2044.2004.03976.x. PMID 15549987
- [Background] Agarwal A, Sinha PK, Tandon M, Dhiraaj S, Singh U. Evaluating the efficacy of the valsalva maneuver on venous cannulation pain: a prospective, randomized study. Anesth Analg. 2005 Oct;101(4):1230-1232. doi: 10.1213/01.ane.0000167270.15047.49. PMID 16192551
- [Background] Cigdem UK, Sevinc S, Esef B, Sureyya O, Muzaffer G, Akif D. [A comparison of three different needles used for spinal anesthesia in terms of squamous epithelial cell transport risk]. Rev Bras Anestesiol. 2017 Sep-Oct;67(5):468-471. doi: 10.1016/j.bjan.2017.04.011. Epub 2017 May 16. Portuguese. PMID 28526468
- [Background] Pstras L, Thomaseth K, Waniewski J, Balzani I, Bellavere F. The Valsalva manoeuvre: physiology and clinical examples. Acta Physiol (Oxf). 2016 Jun;217(2):103-19. doi: 10.1111/apha.12639. Epub 2016 Jan 5. PMID 26662857
- [Background] Macfie AG, Brimacombe J. Response to the Valsalva manoeuvre after spinal anaesthesia. Anaesthesia. 1992 Jan;47(1):13-6. doi: 10.1111/j.1365-2044.1992.tb01944.x. PMID 1536394
- [Background] Looga R. The Valsalva manoeuvre--cardiovascular effects and performance technique: a critical review. Respir Physiol Neurobiol. 2005 May 12;147(1):39-49. doi: 10.1016/j.resp.2005.01.003. PMID 15848122